CLINICAL TRIAL: NCT06048809
Title: A Randomised, Controlled, Examiner Blind, Methodology Development Study to Evaluate the Effect of a Stannous Fluoride Toothpaste on the Oral Microbiome
Brief Title: A Study to Evaluate the Effect of a Stannous Fluoride Toothpaste on the Oral Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 300101
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Results first posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Oral Health

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Toothpaste (Experimental): Participants will be instructed to brush their teeth with the test toothpaste (Sensodyne Repair and Protect containing 1100 parts per million [ppm] fluoride as SnF2) for 1-timed minute twice a day (morning and evening) in their usual manner for 6 weeks. Participants will record each brushing in the diary provided.
  Interventions: Other: Stannous Fluoride Toothpaste (Sensodyne Repair and Protect)
- Reference Toothpaste (Active Comparator): Participants will be instructed to brush their teeth with the reference toothpaste (Colgate Cavity Protection containing 1100 ppm fluoride as sodium monofluorophosphate [SMFP]) for 1-timed minute twice a day (morning and evening) in their usual manner for 6 weeks. Participants will record each brushing in the diary provided.
  Interventions: Other: Regular Fluoride Toothpaste (Colgate Cavity Protection)

INTERVENTIONS:
Other: Stannous Fluoride Toothpaste (Sensodyne Repair and Protect) — Sensodyne Repair and Protect toothpaste containing 1100 ppm fluoride as SnF2.
  Arms: Test Toothpaste
Other: Regular Fluoride Toothpaste (Colgate Cavity Protection) — Colgate Cavity Protection containing 1100 ppm fluoride as SMFP.
  Arms: Reference Toothpaste

SUMMARY:
The aim of this study is to evaluate the effect of a toothpaste containing stannous fluoride (SnF2) over time on the oral bacterial composition and activity and to explore its effect in comparison to a regular fluoride toothpaste.

DETAILED DESCRIPTION:
This will be a single-center, 6-week, randomized, controlled, analyst and examiner-blind, two treatment, parallel group design, methodology development clinical study, investigating the efficacy of a toothpaste containing 0.454 percent (%) SnF2 in healthy adult participants with mild-moderate gingivitis. The study will describe and compare the overall oral bacterial composition and activity following 6 weeks use of a 0.454 % SnF2 toothpaste and regular fluoride toothpaste (control) using microbial and functional profiling techniques. Participants will be instructed to brush twice daily (morning and evening) in their usual manner, for 1-timed minute, for 6 weeks and to record each brushing in the diary provided. Sufficient participants will be screened to ensure approximately 50 participants complete the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant is male or female who, at the time of screening, is aged 18-65 years, inclusive.
* Participant who is willing and able to comply with scheduled visits, sampling schedule, treatment plan and other study procedures.
* Participant, in the opinion of the investigator or medically qualified designee, in good general and mental health.

At Screening (Visit 1):

* Participant with at least 20 natural, permanent teeth (excluding 3rd molars).
* Participant with at least 40 evaluable surfaces.
* Overall mean Turesky Modified Quigley and Hein Plaque Index (TPI) score greater than or equal to (>=) 1.5.
* Participants with 10% less than (<) bleeding sites (BS) < 30%

Exclusion Criteria:

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or otherwise supervised by the investigator, or a member of their immediate family; or a sponsor employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) in the 30 days prior to study entry and/or who is participating in other studies during study participation.
* A participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A participant with any medical/oral condition which, in the opinion of the investigator or medically qualified designee, could impact study outcomes (for example, oral dryness or could directly influence gingival bleeding).
* A participant taking daily doses of medication/having daily treatments which, in the opinion of the investigator or medically qualified designee, could impact study outcomes (for example, is causing oral dryness).
* A participant who is pregnant (self-reported; no pregnancy test required) or intending to become pregnant over the course of the study.
* A participant who is breastfeeding.
* A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* A participant who is unwilling or unable to comply with the Lifestyle Considerations described in this protocol.
* A participant who has difficulty complying with study procedures and examinations, such as excessive gagging during oral assessments.
* A participant who has had routine dental prophylaxis within 12 weeks of Screening.
* A participant who has undergone a tooth bleaching procedure (at-home or professional) within 8 weeks of Screening.
* A participant with any of the following which, in the opinion of the investigator or medically qualified designee, could impact study outcomes or the oral health of the participants if they were to participate in the study:

  1. Severe gingivitis.
  2. Signs of active periodontal disease or who is receiving or has received treatment for periodontal disease (including surgery) within 12 months of Screening.
  3. Active caries.
  4. Evidence of gross intra-oral neglect or the need for extensive dental therapy.
  5. Restorations in a poor state of repair or metal fillings.
  6. Any dental condition (example, malalignment, overcrowding)
  7. High levels of extrinsic dental stain or calculus deposits.
* A participant with the following:

  1. A tongue or lip piercing.
  2. Multiple dental implants which, in the opinion of the investigator or medically qualified designee, could impact study outcomes.
  3. Fixed bridge(s) or removable partial dentures.
  4. Has or has had fixed or removable orthodontic braces/bands or a fixed orthodontic retainer within 3 months of Screening.
* A participant who is unwilling to forgo use of an orthodontic retainer for the duration of the study, provided there would be no impact on the outcome of any previous, completed orthodontic treatment or the participant's well-being.
* Participant who is a current smoker or an ex-smoker who stopped within 6 months of Screening (Visit 1).
* Participant who is a currently user of recreational drugs (example, cannabis) within 6 months of Screening.
* Participant who currently uses smokeless forms of tobacco (example, chewing tobacco, nicotine-based e-cigarettes) within 6 months of Screening.
* Visit 1 (Screening)

  1. A participant who has taken antibiotics within 4 weeks of Screening.
  2. Participant who has used an anti-bacterial mouthwash (example, chlorhexidine) or another oral care product within 2 weeks of Screening that, in the opinion of the investigator or dentally qualified designee, could affect plaque formation or gingival health.
* Visit 2 (Baseline)

  1. A participant who has taken antibiotics during the lead-in period (between Screening and Baseline).
* Participant with a recent history (within the last year) of alcohol or other substance abuse.
* A participant who has previously been enrolled in this study.
* Participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Salus Research, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in the United States.
Pre-assignment Details: A total of 59 participants were screened of which 56 participants were enrolled, and 55 participants were randomized to receive treatment in 2 groups: Test Product group (28 participants) and Reference Product group (27 participants). 4 screened participants were not randomized (3 participants did not meet the study criteria and 1 participant was lost to follow-up). A total of 51 randomized participants completed the study.
Groups:
- Test Product (Sensodyne Repair and Protect): Participants were instructed to apply a ribbon of test product (Sensodyne Repair and Protect toothpaste) containing 1100 parts per million [ppm] fluoride as stannous fluoride (SnF2) across the full brush head of toothbrush provided and brush their teeth for one timed minute twice daily (morning and evening) in their usual manner for 6 weeks.
- Reference Product (Colgate Cavity Protection): Participants were instructed to apply a ribbon of reference product (Colgate Cavity Protection toothpaste) containing 1100 ppm fluoride as sodium monofluorophosphate [SMFP] across the full brush head of toothbrush provided and brush their teeth for one timed minute twice daily (morning and evening) in their usual manner for 6 weeks.
Period: Overall Study
Arm/Group | Test Product (Sensodyne Repair and Protect) | Reference Product (Colgate Cavity Protection)
Started | 28 | 27
Completed | 25 | 26
Not Completed | 3 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who completed at least one use of study product.
Groups:
- Test Product (Sensodyne Repair and Protect): Participants were instructed to apply a ribbon of test product (Sensodyne Repair and Protect toothpaste) containing 1100 ppm fluoride as SnF2 across the full brush head of toothbrush provided and brush their teeth for one timed minute twice daily (morning and evening) in their usual manner for 6 weeks.
- Reference Product (Colgate Cavity Protection): Participants were instructed to apply a ribbon of reference product (Colgate Cavity Protection toothpaste) containing 1100 ppm fluoride as SMFP across the full brush head of toothbrush provided and brush their teeth for one timed minute twice daily (morning and evening) in their usual manner for 6 weeks.
- Total: Total of all reporting groups
Arm/Group | Test Product (Sensodyne Repair and Protect) | Reference Product (Colgate Cavity Protection) | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (12.11) | 46.2 (10.85) | 44.2 (11.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 24 | 27 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 4 | 0 | 4
  Asian - Central/South Asian Heritage | 1 | 0 | 1
  White - Arabic/North African Heritage | 0 | 1 | 1
  White - White/Caucasian/European Heritage | 22 | 26 | 48
  Multiple | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Alpha Diversity at Baseline (Day 1)
Description: Alpha diversity was defined as species diversity in sites or habitats and was used to describe the overall oral bacterial composition. Samples were collected from 4 different areas of mouth (tongue, supragingival plaque, subgingival surface, and saliva) and microbial profiling (16S ribosomal ribonucleic acid [rRNA] gene amplicon analysis) was performed to identify the bacteria present within a given sample down to the genus and/or species level. Alpha diversity (overall) was measured using Shannon index. Shannon Index was derived as the negative of the sum of the p*ln(p) across all species in the sample where p was the proportion of the sample made up from each species. Index scores ranged from 0 to ln(S) where S was the number of species in the sample. Higher values indicated greater diversity and a more complex community with a more even distribution of species. Lower values indicated lower diversity, suggesting dominance by a few species or a less complex community.
Time Frame: Baseline (Day 1)
Population: Microbiome Population included all randomized participants who completed at least one use of the study product and had an evaluable microbiome result (at least one area at both Baseline and Week 6).
Measure: Median (Inter-Quartile Range); unit: Shannon index
Arm/Group | Test Product (Sensodyne Repair and Protect) | Reference Product (Colgate Cavity Protection)
Number analyzed (Participants) | 25 | 26
Shannon index | 3.7 [3.3 to 3.9] | 3.5 [3.1 to 3.9]

2. Primary Outcome: Alpha Diversity at Week 6
Description: Alpha diversity was defined as species diversity in sites or habitats and was used to describe the overall oral bacterial composition. Samples were collected from 4 different areas of mouth (tongue, supragingival plaque, subgingival surface, and saliva) and microbial profiling (16S rRNA gene amplicon analysis) was performed to identify the bacteria present within a given sample down to the genus and/or species level. Alpha diversity (overall) was measured using Shannon index. Shannon Index was derived as the negative of the sum of the p*ln(p) across all species in the sample where p was the proportion of the sample made up from each species. Index scores ranged from 0 to ln(S) where S was the number of species in the sample. Higher values indicated greater diversity and a more complex community with a more even distribution of species. Lower values indicated lower diversity, suggesting dominance by a few species or a less complex community.
Time Frame: Week 6
Population: Microbiome Population.
Measure: Median (Inter-Quartile Range); unit: Shannon index
Arm/Group | Test Product (Sensodyne Repair and Protect) | Reference Product (Colgate Cavity Protection)
Number analyzed (Participants) | 25 | 26
Shannon index | 3.8 [3.3 to 4.0] | 3.6 [3.2 to 4.0]

3. Primary Outcome: Adjusted Mean Change From Baseline in Abundance for Each Bacterial Group Assessed by Differential Abundance Analysis at Week 6 (Test Product)
Description: Analysis of Compositions of Microbiomes with Bias Correction, version 2 (ANCOM-BC2) method was used to identify bacterial species that were differentially abundant between Baseline and Week 6. Samples were collected from 4 different areas of mouth (tongue, supragingival plaque, subgingival surface, and saliva) at the indicated timepoints, and differential abundance analysis was performed. Change from Baseline was calculated by subtracting the Baseline value from the value at Week 6. Baseline was defined as Day 1. Log-fold change from Baseline in abundance (overall) for each bacterial group was reported.
Time Frame: Baseline and Week 6
Population: Microbiome Population.
Measure: Mean (Standard Error); unit: log fold change
Groups:
- Test Product (Sensodyne Repair and Protect Toothpaste): Participants were instructed to apply a ribbon of test product (Sensodyne Repair and Protect toothpaste) containing 1100 ppm fluoride as SnF2 across the full brush head of toothbrush provided and brush their teeth for one timed minute twice daily (morning and evening) in their usual manner for 6 weeks.
Arm/Group | Test Product (Sensodyne Repair and Protect Toothpaste)
Number analyzed (Participants) | 25
log fold change
  Haemophilus parainfluenzae | -1.44299 (0.341277)
  Neisseria elongata | -1.15069 (0.391919)
  Aggregatibacter species (sp.)_Human Microbial Taxon (HMT)_898 | -1.00158 (0.356817)
  Parvimonas sp._HMT_110 | -1.04854 (0.386699)
  Aggregatibacter aphrophilus | -0.99362 (0.3691)
  Kingella oralis | -1.09495 (0.409102)
  Haemophilus sp._HMT_036 | -0.89269 (0.364569)
  Haemophilus haemolyticus | -0.94098 (0.403023)
  Neisseria mucosa | -0.77591 (0.333405)
  Parvimonas sp._HMT_393_nov_97.053 percent (%) | -0.95005 (0.411073)
  Ottowia sp._HMT_894 | -0.74756 (0.3261)
  Cryptobacterium curtum | 0.75985 (0.334759)
  Lautropia mirabilis | -0.92156 (0.408231)
  Haemophilus paraphrohaemolyticus | -0.68962 (0.307868)
  Capnocytophaga sp._HMT_332 | -0.68115 (0.306965)
  Neisseria flavescens | -1.11659 (0.509096)
  Capnocytophaga gingivalis_nov_96.429% | -0.72364 (0.34236)
  Capnocytophaga sputigena | -0.83191 (0.399852)
  Haemophilus sputorum | -0.81061 (0.390197)
  Capnocytophaga gingivalis_nov_90.546% | -0.64962 (0.313955)
  Prevotella denticola | 0.908887 (0.458641)
  Aggregatibacter sp._HMT_513 | -0.81317 (0.418317)
  Veillonella sp._HMT_780 | -0.62127 (0.323856)
  Neisseria perflava | -0.98271 (0.519658)
  Slackia exigua | 0.61058 (0.333686)
  Shuttleworthia satelles | 0.615042 (0.34007)
  Aggregatibacter sp._HMT_458 | -0.75679 (0.423703)
  Ruminococcaceae_[G-1] bacterium_HMT_075 | 0.752979 (0.421849)
  Campylobacter showae | -0.77501 (0.440186)
  Streptococcus sp._HMT_056 | -0.62733 (0.36379)
Statistical Analysis 1: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Haemophilus parainfluenzae: Change From Baseline at Week 6; Test type: Other; p = 0.0000236, ANCOM-BC2
Statistical Analysis 2: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Neisseria elongata: Change From Baseline at Week 6; Test type: Other; p = 0.0033243, ANCOM-BC2
Statistical Analysis 3: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Aggregatibacter sp._HMT_898: Change From Baseline at Week 6; Test type: Other; p = 0.00500088, ANCOM-BC2
Statistical Analysis 4: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Parvimonas sp._HMT_110: Change From Baseline at Week 6; Test type: Other; p = 0.0066975, ANCOM-BC2
Statistical Analysis 5: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Aggregatibacter aphrophilus: Change From Baseline at Week 6; Test type: Other; p = 0.00710228, ANCOM-BC2
Statistical Analysis 6: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Kingella oralis: Change From Baseline at Week 6; Test type: Other; p = 0.00744022, ANCOM-BC2
Statistical Analysis 7: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Haemophilus sp._HMT_036: Change From Baseline at Week 6; Test type: Other; p = 0.01434037, ANCOM-BC2
Statistical Analysis 8: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Haemophilus haemolyticus: Change From Baseline at Week 6; Test type: Other; p = 0.01955327, ANCOM-BC2
Statistical Analysis 9: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Neisseria mucosa: Change From Baseline at Week 6; Test type: Other; p = 0.01995277, ANCOM-BC2
Statistical Analysis 10: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Parvimonas sp._HMT_393_nov_97.053%: Change From Baseline at Week 6; Test type: Other; p = 0.02082528, ANCOM-BC2
Statistical Analysis 11: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Ottowia sp._HMT_894: Change from Baseline at Week 6; Test type: Other; p = 0.02188156, ANCOM-BC2
Statistical Analysis 12: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Cryptobacterium curtum: Change From Baseline at Week 6; Test type: Other; p = 0.02321733, ANCOM-BC2
Statistical Analysis 13: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Lautropia mirabilis: Change from Baseline at Week 6; Test type: Other; p = 0.02397996, ANCOM-BC2
Statistical Analysis 14: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Haemophilus paraphrohaemolyticus: Change From Baseline at Week 6; Test type: Other; p = 0.02509094, ANCOM-BC2
Statistical Analysis 15: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Capnocytophaga sp._HMT_332: Change From Baseline at Week 6; Test type: Other; p = 0.02648847, ANCOM-BC2
Statistical Analysis 16: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Neisseria flavescens: Change From Baseline at Week 6; Test type: Other; p = 0.02828764, ANCOM-BC2
Statistical Analysis 17: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Capnocytophaga gingivalis_nov_96.429%: Change From Baseline at Week 6; Test type: Other; p = 0.03454372, ANCOM-BC2
Statistical Analysis 18: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Capnocytophaga sputigena: Change From Baseline at Week 6; Test type: Other; p = 0.03747507, ANCOM-BC2
Statistical Analysis 19: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Haemophilus sputorum: Change From Baseline at Week 6; Test type: Other; p = 0.03776136, ANCOM-BC2
Statistical Analysis 20: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Capnocytophaga gingivalis_nov_90.546%: Change From Baseline at Week 6; Test type: Other; p = 0.03853215, ANCOM-BC2
Statistical Analysis 21: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Prevotella denticola: Change From Baseline at Week 6; Test type: Other; p = 0.04751303, ANCOM-BC2
Statistical Analysis 22: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Aggregatibacter sp._HMT_513: Change From Baseline at Week 6; Test type: Other; p = 0.05190512, ANCOM-BC2
Statistical Analysis 23: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Veillonella sp._HMT_780: Change From Baseline at Week 6; Test type: Other; p = 0.0550647, ANCOM-BC2
Statistical Analysis 24: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Neisseria perflava: Change From Baseline at Week 6; Test type: Other; p = 0.05861488, ANCOM-BC2
Statistical Analysis 25: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Slackia exigua: Change From Baseline at Week 6; Test type: Other; p = 0.06727926, ANCOM-BC2
Statistical Analysis 26: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Shuttleworthia satelles: Change from Baseline at Week 6; Test type: Other; p = 0.07051698, ANCOM-BC2
Statistical Analysis 27: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Aggregatibacter sp._HMT_458: Change From Baseline at Week 6; Test type: Other; p = 0.0740793, ANCOM-BC2
Statistical Analysis 28: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Ruminococcaceae_[G-1] bacterium_HMT_075: Change From Baseline at Week 6; Test type: Other; p = 0.07426973, ANCOM-BC2
Statistical Analysis 29: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Campylobacter showae: Change From Baseline at Week 6; Test type: Other; p = 0.07829888, ANCOM-BC2
Statistical Analysis 30: Comparison: Test Product (Sensodyne Repair and Protect Toothpaste); Streptococcus sp._HMT_056: Change From Baseline at Week 6; Test type: Other; p = 0.08462924, ANCOM-BC2

4. Primary Outcome: Adjusted Mean Change From Baseline in Abundance for Each Bacterial Group Assessed by Differential Abundance Analysis at Week 6 (Reference Product)
Description: ANCOM-BC2 method was used to identify bacterial species that were differentially abundant between Baseline and Week 6. Samples were collected from 4 different areas of mouth (tongue, supragingival plaque, subgingival surface, and saliva) at the indicated timepoints, and differential abundance analysis was performed. Change from Baseline was calculated by subtracting the Baseline value from the value at Week 6. Baseline was defined as Day 1. Log-fold change from Baseline in abundance (overall) for each bacterial group was reported.
Time Frame: Baseline and Week 6
Population: Microbiome Population.
Measure: Mean (Standard Error); unit: log fold change
Arm/Group | Reference Product (Colgate Cavity Protection)
Number analyzed (Participants) | 26
log fold change
  Abiotrophia defectiva | -0.77816 (0.417556)
  Saccharibacteria_(TM7)_[G1] bacterium_HMT_346 | 0.819312 (0.441412)
  Olsenella sp._HMT_807 | 0.742059 (0.409411)
  Fusobacterium nucleatum_nucleatum_subspecies(subsp.)_animalis | 0.725497 (0.414044)
  Bergeyella sp._HMT_322 | -0.45915 (0.274711)
  Peptostreptococcaceae_[XI][G-1] [Eubacterium]_infirmum | 0.529594 (0.318012)
  Prevotella sp._HMT_317 | 0.754675 (0.469454)
  Bacteroidales_[G-2] bacterium_HMT_274 | 0.656014 (0.409449)
  Actinomyces sp._HMT_175_nov 97.951% | -0.575 (0.360622)
  Slackia exigua | 0.476852 (0.307014)
  Granulicatella adiacens | -0.42768 (0.277858)
  Prevotella oris | 0.604954 (0.393279)
  Streptococcus sp._HMT_064 | -0.65561 (0.436817)
  Schaalia odontolyticus | -0.74594 (0.511306)
  Mogibacterium diversum | 0.490377 (0.338375)
  Prevotella denticola | 0.592222 (0.410061)
  Absconditabacteria_(SR1)_[G-1] bacterium_HMT_875 | -0.35571 (0.24693)
  Prevotella nigrescens | 0.57069 (0.400784)
  Streptococcus chosunense | -0.62541 (0.443126)
Statistical Analysis 1: Comparison: Reference Product (Colgate Cavity Protection); Abiotrophia defectiva: Change from Baseline at Week 6; Test type: Other; p = 0.062378, ANCOM-BC2
Statistical Analysis 2: Comparison: Reference Product (Colgate Cavity Protection); Saccharibacteria_(TM7)_[G1] bacterium_HMT_346: Change from Baseline at Week 6; Test type: Other; p = 0.063437, ANCOM-BC2
Statistical Analysis 3: Comparison: Reference Product (Colgate Cavity Protection); Olsenella sp._HMT_807: Change from Baseline at Week 6; Test type: Other; p = 0.069908, ANCOM-BC2
Statistical Analysis 4: Comparison: Reference Product (Colgate Cavity Protection); Fusobacterium nucleatum_nucleatum_subsp._animalis: Change from Baseline at Week 6; Test type: Other; p = 0.079736, ANCOM-BC2
Statistical Analysis 5: Comparison: Reference Product (Colgate Cavity Protection); Bergeyella sp._HMT_322: Change from Baseline at Week 6; Test type: Other; p = 0.094642, ANCOM-BC2
Statistical Analysis 6: Comparison: Reference Product (Colgate Cavity Protection); Peptostreptococcaceae_[XI][G-1] [Eubacterium]_infirmum: Change from Baseline at Week 6; Test type: Other; p = 0.095848, ANCOM-BC2
Statistical Analysis 7: Comparison: Reference Product (Colgate Cavity Protection); Prevotella sp._HMT_317: Change from Baseline at Week 6; Test type: Other; p = 0.107931, ANCOM-BC2
Statistical Analysis 8: Comparison: Reference Product (Colgate Cavity Protection); Bacteroidales_[G-2] bacterium_HMT_274: Change from Baseline at Week 6; Test type: Other; p = 0.109114, ANCOM-BC2
Statistical Analysis 9: Comparison: Reference Product (Colgate Cavity Protection); Actinomyces sp._HMT_175_nov 97.951%: Change from Baseline at Week 6; Test type: Other; p = 0.11083, ANCOM-BC2
Statistical Analysis 10: Comparison: Reference Product (Colgate Cavity Protection); Slackia exigua: Change from Baseline at Week 6; Test type: Other; p = 0.120377, ANCOM-BC2
Statistical Analysis 11: Comparison: Reference Product (Colgate Cavity Protection); Granulicatella adiacens: Change from Baseline at Week 6; Test type: Other; p = 0.123758, ANCOM-BC2
Statistical Analysis 12: Comparison: Reference Product (Colgate Cavity Protection); Prevotella oris: Change from Baseline at Week 6; Test type: Other; p = 0.123992, ANCOM-BC2
Statistical Analysis 13: Comparison: Reference Product (Colgate Cavity Protection); Streptococcus sp._HMT_064: Change from Baseline at Week 6; Test type: Other; p = 0.133385, ANCOM-BC2
Statistical Analysis 14: Comparison: Reference Product (Colgate Cavity Protection); Schaalia odontolyticus: Change from Baseline at Week 6; Test type: Other; p = 0.144598, ANCOM-BC2
Statistical Analysis 15: Comparison: Reference Product (Colgate Cavity Protection); Mogibacterium diversum: Change from Baseline at Week 6; Test type: Other; p = 0.147278, ANCOM-BC2
Statistical Analysis 16: Comparison: Reference Product (Colgate Cavity Protection); Prevotella denticola: Change from Baseline at Week 6; Test type: Other; p = 0.148674, ANCOM-BC2
Statistical Analysis 17: Comparison: Reference Product (Colgate Cavity Protection); Absconditabacteria_(SR1)_[G-1] bacterium_HMT_875: Change from Baseline at Week 6; Test type: Other; p = 0.149722, ANCOM-BC2
Statistical Analysis 18: Comparison: Reference Product (Colgate Cavity Protection); Prevotella nigrescens: Change from Baseline at Week 6; Test type: Other; p = 0.154465, ANCOM-BC2
Statistical Analysis 19: Comparison: Reference Product (Colgate Cavity Protection); Streptococcus chosunense: Change from Baseline at Week 6; Test type: Other; p = 0.158139, ANCOM-BC2

ADVERSE EVENTS:
Time Frame: From signing of informed consent form until 5 days after last administration of study product or last study procedure (up to approximately 51 days)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study product including any washout or lead-in product (or medical device), whether or not considered related to the study product, including any washout or lead-in product (or medical device). A Serious Adverse Event (SAE) was a particular category of an AE where the adverse outcome is serious.
Arm/Group | Test Product (Sensodyne Repair and Protect) | Reference Product (Colgate Cavity Protection)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 3/28 | 0/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product (Sensodyne Repair and Protect) (N=28) | Reference Product (Colgate Cavity Protection) (N=27)
APHTHOUS ULCER (Gastrointestinal disorders) | 1 | 0
ORAL MUCOSAL EXFOLIATION (Gastrointestinal disorders) | 1 | 0
TONGUE EXFOLIATION (Gastrointestinal disorders) | 1 | 0
SUNSCREEN SENSITIVITY (Immune system disorders) | 1 | 0
PERIORAL DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/09/NCT06048809/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT06048809/SAP_001.pdf